CLINICAL TRIAL: NCT02642393
Title: A Randomized, Double-blind, Placebo-controlled Trial of Urate-elevating Inosine Treatment to Slow Clinical Decline in Early Parkinson's Disease
Brief Title: Study of Urate Elevation in Parkinson's Disease, Phase 3
Acronym: SURE-PD3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Michael Alan Schwarzschild (Other)
Collaborators: The Parkinson Study Group (Network); Michael J. Fox Foundation for Parkinson's Research (Other); University of Rochester (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Michael Alan Schwarzschild, Chair, SURE-PD3 Steering Committee, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: INO-PD-P3-2014; 1U01NS090259-01A1 (NIH)
Record Dates: First submitted 2015-12-19; First posted 2015-12-30 (Estimated); Results first posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Parkinson's Disease
Keywords: SURE-PD3; Parkinson's disease; PD; Inosine; Urate; Parkinson Study Group (PSG)
MeSH Terms: conditions — Parkinson Disease | interventions — Inosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inosine (Experimental): Inosine will be dosed by titrating the number of capsules taken daily to achieve an elevation of serum urate to trough levels of 7.1 to 8.0 mg/dL.
  Interventions: Drug: Inosine
- Placebo (Placebo Comparator): Placebo will be dosed to match the capsule titrations of the inosine group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inosine — capsules containing 500 mg of inosine
  Other Names: hypoxanthine 9-β-D-ribofuranoside
  Arms: Inosine
Drug: Placebo — capsules containing ~500 mg of lactose and appearing indistinguishable from inosine capsules
  Other Names: inactive agent
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled, phase 3 trial to determine whether oral inosine dosed to moderately elevate serum urate (from ≤5.7 mg/dL to 7.1-8.0 mg/dL) over 2 years slows clinical decline in early PD.

Clinical decline will be assessed as change in the primary outcome variable of the Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS), a composite scale comprising patient- and clinician-reported outcomes.

DETAILED DESCRIPTION:
Capsules containing 500 mg of inosine (active drug) or ~500 mg of lactose (placebo) will be taken orally up to two capsules three times per day (i.e., up to 3 g/day) for 24 months. In the inosine-treated group the number of capsules taken per day will be titrated to serum urate levels - measured at trough at study visits no more than three months apart - in order to achieve concentrations of 7.1-8.0 mg/dL. Initial dosing will be tailored to individualized factors including gender and pretreatment serum urate, and then advanced gradually toward the projected target dose. Adjustments in dosing of placebo capsules in the control arm will be algorithm-based to match dosing of inosine capsules in the active drug arm.

Following study drug discontinuation all subjects will be followed during a 3-month wash-out period by telephone calls and a final study visit. All study visits after screening will include measurement of the primary outcome variable (MDS-UPDRS) and most will include secondary outcome variables: adverse events, dose adjustments, disability warranting initiation of dopaminergic therapy, Quality of Life in Neurological Disorders (Neuro-QOL), 39-item Parkinson's Disease Questionnaire (PDQ-39), Schwab & England Activities of Daily Living (S&E ADL) scale, Montreal Cognitive Assessment (MoCA), and orthostatic vital signs.

ELIGIBILITY:
INCLUSION CRITERIA:

Study subjects meeting all of the following criteria will be allowed to enroll in the study:

1. Willingness and ability to give written informed consent and to comply with trial procedures.
2. Fulfillment of diagnostic criteria for idiopathic PD with at least two of the cardinal signs of PD (resting tremor, bradykinesia, rigidity) present at 2nd screening and baseline evaluations, as assessed by the Site Investigator.
3. Absence of current or imminent (within 90 days of enrollment) PD disability requiring dopaminergic therapy, as assessed by the Site Investigator.
4. Modified Hoehn and Yahr Scale Stage 1 to 2.5 inclusive.
5. Age 30 or older at the time of PD diagnosis.
6. Diagnosis of PD made within 3 years prior to 1st Screening Visit.
7. Non-fasting serum urate ≤ 5.7 mg/dL at 1st Screening Visit (SC1).
8. If the subject is female, then:

   1. Being surgically sterile (hysterectomy or tubal ligation), or
   2. Being postmenopausal (last menstruation was two years or more prior to 2nd Screening Visit), or
   3. For those of childbearing potential

      * Using a reliable form of contraception for 60 days or more prior to Baseline Visit and agreeing to continue such use for 30 days post last dose of study drug. Reliable forms of contraception include: abstinence; implanted, injected or oral contraceptives (birth control pills), intrauterine device in place for at least 3 months prior to Baseline Visit, vaginal ring with spermicide, barrier with spermicide such as male or female condom, diaphragm or cervical cap, transdermal patch; male partner with vasectomy.
      * And having a negative pregnancy test at the 2nd Screening Visit. [Note that a urine pregnancy test will be performed at screening on all women who are not at least two years postmenopausal or surgically sterile.]

EXCLUSION CRITERIA:

Study subjects meeting any of the following criteria during screening evaluations will be excluded from entry into the study:

1. Atypical parkinsonism, including that due to drugs, metabolic disorders, encephalitis, cerebrovascular disease, normal pressure hydrocephalus, or other neurodegenerative disease.
2. Dopamine transporter (DAT) brain scan without evidence of dopamine deficit.
3. History of gout.
4. History of uric acid or urate urolithiasis, or recurrent urolithiasis all of unknown type.
5. A screening test positive for uric acid crystalluria, urine pH ≤ 5.0, or an estimated glomerular filtration rate < 60 ml/min/1.73 m2.
6. History of myocardial infarction or stroke.
7. Symptomatic congestive heart failure with a documented ejection fraction below 45%.
8. History of severe chronic obstructive pulmonary disease.
9. Mini Mental State Exam score < 25; i.e., a score of 0 to 24.
10. Use of any anti-parkinsonian medication (including levodopa, dopamine agonists, amantadine, entacapone and the anticholinergic agents trihexyphenidyl and benztropine) other than monoamine oxidase-B inhibitors within 60 days of Baseline, or in excess of 90 days.
11. Change in the dosage of (or initiation of) a monoamine oxidase-B (MAO-B) inhibitor within 90 days prior to Baseline, i.e., entry on a MAO-B inhibitor requires a stable dosage for the 90 days prior to Baseline.
12. Use of the following within 30 days prior to the Baseline Visit: inosine, allopurinol, febuxostat, probenecid, more than 50 IU of vitamin E daily, or more than 300 mg of vitamin C daily (though a daily standard multivitamin such as Bayer One-A-Day® or Centrum® is permissible), reserpine, methylphenidate, amphetamines, cinnarizine, monoamine oxidase-A inhibitors, tetrabenazine, neuroleptics or other dopamine blocking drugs.
13. Use of the following within 90 days prior to the DAT neuroimaging screening evaluation: modafinil, armodafinil, metoclopramide, alpha-methyldopa, methylphenidate, reserpine, or amphetamine derivative.
14. Unstable dosing of a thiazide -- such as hydrochlorothiazide (e.g., Esidrex), chlorothiazide (e.g., Diuril), chlorthalidone (e.g., Hygroton), indapamide (e.g., Lozol), metolazone (e.g., Zaroxolyn), which are permissible as long as the subject is on a stable dose from 1 week prior to the 1st Screening Visit through the Baseline Visit.
15. Known unstable medical or psychiatric condition that may compromise participation in the study. (Note that difficulty swallowing large capsules might preclude participation due to the size of the study drug capsules.)
16. Clinically serious abnormality in the screening visit laboratory studies or ECG, as determined by the Site Investigator.
17. Participation in another investigational treatment study within 30 days prior to the Baseline Visit.
18. Known hypersensitivity or intolerability to inosine.
19. Known hypersensitivity to DaTscan (either the active substance of ioflupane I-123 or to any of the excipients).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Schwarzschild, MD, PhD, Study Chair — Massachusetts General Hospital (PI of Clinical Coordinating Center), PSG (Chair, SURE-PD3 Steering Committee); Alberto Ascherio, MD, DrPH, Study Director — Harvard School of Public Health, PSG (Co-Chair, SURE-PD3 Steering Committee); David Oakes, PhD, Study Director — University of Rochester (PI of Data Coordinating Center), PSG (Study Statistician/Member, SURE-PD3 Steering Committee); Eric A Macklin, PhD, Study Director — Massachusetts General Hospital, PSG (Study Statistician/Member, SURE-PD3 Steering Committee)
Locations (62):
- United States (61):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of California San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California Davis, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Rocky Mountain Movement Disorder Center, Englewood, Colorado
  - Hartford HealthCare Movement Disorders Center, Vernon, Connecticut
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Neurosciences Institute at Central DuPage Hospital, Winfield, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Oschner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Henry Ford Health System, West Bloomfield, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Overlook Medical Center, Atlantic Neuroscience Institute, Summit, New Jersey
  - Albany Medical College, Albany, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Weill Cornell Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke University, Durham, North Carolina
  - University of Cincinnati/Cincinnati Children's Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Wesley Neurology Clinic, PC, Cordova, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Houston Medical School, Houston, Texas
  - Baylor Scott & White Health, Temple, Texas
  - The University of Vermont, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - VCU Parkinson's & Movement Disorder Center (McGuire Veterans Hospital), Richmond, Virginia
  - Sentara Neurology Specialists, Virginia Beach, Virginia
  - Inland Northwest Research, Spokane, Washington
  - Northwest Neurological PLLC, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- University of Puerto Rico, San Juan, Massachusetts, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
De-identified data; per policies of NIH/NINDS and the PSG (Parkinson Study Group)

REFERENCES:
- [Background] Parkinson Study Group SURE-PD Investigators; Schwarzschild MA, Ascherio A, Beal MF, Cudkowicz ME, Curhan GC, Hare JM, Hooper DC, Kieburtz KD, Macklin EA, Oakes D, Rudolph A, Shoulson I, Tennis MK, Espay AJ, Gartner M, Hung A, Bwala G, Lenehan R, Encarnacion E, Ainslie M, Castillo R, Togasaki D, Barles G, Friedman JH, Niles L, Carter JH, Murray M, Goetz CG, Jaglin J, Ahmed A, Russell DS, Cotto C, Goudreau JL, Russell D, Parashos SA, Ede P, Saint-Hilaire MH, Thomas CA, James R, Stacy MA, Johnson J, Gauger L, Antonelle de Marcaida J, Thurlow S, Isaacson SH, Carvajal L, Rao J, Cook M, Hope-Porche C, McClurg L, Grasso DL, Logan R, Orme C, Ross T, Brocht AF, Constantinescu R, Sharma S, Venuto C, Weber J, Eaton K. Inosine to increase serum and cerebrospinal fluid urate in Parkinson disease: a randomized clinical trial. JAMA Neurol. 2014 Feb;71(2):141-50. doi: 10.1001/jamaneurol.2013.5528. PMID 24366103
- [Derived] Di Luca DG, Macklin EA, Hodgeman K, Lopez G, Pothier L, Callahan KF, Lowell J, Chan J, Videnovic A, Lungu C, Lang AE, Litvan I, Schwarzschild MA, Simuni T. Enrollment of Participants From Marginalized Racial and Ethnic Groups: A Comparative Assessment of the STEADY-PD III and SURE-PD3 Trials. Neurol Clin Pract. 2023 Feb;13(1):e200113. doi: 10.1212/CPJ.0000000000200113. Epub 2023 Jan 18. PMID 36865634
- [Derived] Parkinson Study Group SURE-PD3 Investigators; Schwarzschild MA, Ascherio A, Casaceli C, Curhan GC, Fitzgerald R, Kamp C, Lungu C, Macklin EA, Marek K, Mozaffarian D, Oakes D, Rudolph A, Shoulson I, Videnovic A, Scott B, Gauger L, Aldred J, Bixby M, Ciccarello J, Gunzler SA, Henchcliffe C, Brodsky M, Keith K, Hauser RA, Goetz C, LeDoux MS, Hinson V, Kumar R, Espay AJ, Jimenez-Shahed J, Hunter C, Christine C, Daley A, Leehey M, de Marcaida JA, Friedman JH, Hung A, Bwala G, Litvan I, Simon DK, Simuni T, Poon C, Schiess MC, Chou K, Park A, Bhatti D, Peterson C, Criswell SR, Rosenthal L, Durphy J, Shill HA, Mehta SH, Ahmed A, Deik AF, Fang JY, Stover N, Zhang L, Dewey RB Jr, Gerald A, Boyd JT, Houston E, Suski V, Mosovsky S, Cloud L, Shah BB, Saint-Hilaire M, James R, Zauber SE, Reich S, Shprecher D, Pahwa R, Langhammer A, LaFaver K, LeWitt PA, Kaminski P, Goudreau J, Russell D, Houghton DJ, Laroche A, Thomas K, McGraw M, Mari Z, Serrano C, Blindauer K, Rabin M, Kurlan R, Morgan JC, Soileau M, Ainslie M, Bodis-Wollner I, Schneider RB, Waters C, Ratel AS, Beck CA, Bolger P, Callahan KF, Crotty GF, Klements D, Kostrzebski M, McMahon GM, Pothier L, Waikar SS, Lang A, Mestre T. Effect of Urate-Elevating Inosine on Early Parkinson Disease Progression: The SURE-PD3 Randomized Clinical Trial. JAMA. 2021 Sep 14;326(10):926-939. doi: 10.1001/jama.2021.10207. PMID 34519802
- [Derived] Mestre TA, Macklin EA, Ascherio A, Ferreira JJ, Lang AE, Schwarzschild MA; Parkinson Study Group SURE-PD3 Investigators. Expectations of Benefit in a Trial of a Candidate Disease-Modifying Treatment for Parkinson Disease. Mov Disord. 2021 Aug;36(8):1964-1967. doi: 10.1002/mds.28630. Epub 2021 May 4. PMID 33942376
- See also: Not-for-profit scientific network of Parkinson centers in North America — http://www.parkinson-study-group.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inosine | Placebo
Started | 149 | 149
Completed | 50 (Participants who completed the study: On-drug: 31; In-person off-drug:13; By telephone off-drug: 6) | 57 (Participants who completed the study: On-drug: 40; In-person off-drug: 16; By telephone off-drug: 1)
Not Completed | 99 | 92

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inosine | Placebo | Total
Number analyzed (Participants) | 149 | 149 | 298
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 76 | 75 | 151
  >=65 years | 73 | 74 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (9.7) | 63.6 (9.4) | 63.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 67 | 147
  Male | 69 | 82 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 144 | 145 | 289
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 143 | 145 | 288
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 1 | 0 | 1
  United States | 148 | 149 | 297

OUTCOME MEASURES:

1. Primary Outcome: Rate of Clinical Decline
Description: The primary outcome of the trial is rate of change in the Movement Disorders Society Unified PD Rating Scale (MDS-UPDRS) I-III total score over 24 months estimated from a shared-baseline, random-slopes mixed model, censoring follow-up of subjects after initiation of dopaminergic therapy. Parts I-III of the MDS-UPDRS include ratings of non-motor experiences of daily living, motor experiences of daily living, and a motor examination. The MDS-UPDRS is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse symptoms. Parts I-III contain 59 total questions (13 in Part I, 13 in Part II, and 33 in Part III). Total scores for Parts I-III are calculated as simple sums of component items with mean imputation by Part if no more than 1, 2, or 7 items are missing for Parts I through III, respectively. Total scores may range from 0 to 236, with 0 meaning no symptoms and 236 meaning worse symptoms.
Time Frame: two years
Measure: Mean (95% Confidence Interval); unit: score per year
Arm/Group | Inosine | Placebo
Number analyzed (Participants) | 149 | 149
score per year | 11.116 [9.669 to 12.563] | 9.860 [8.410 to 11.310]
Statistical Analysis 1: Comparison: Inosine vs Placebo; Test type: Other; p = 0.183, Mixed Models Analysis; Slope = 1.256, 95% CI 2-sided [-0.594 to 3.106], Standard Error of Mean 0.943

2. Secondary Outcome: Rate of Developing Adverse Effects
Description: Safety also will be evaluated by comparing active vs. placebo treatment with respect to overall adverse event (AE) and serious AE (SAE) rate.
Time Frame: two years
Population: Only 147 of 149 participants in the inosine group were analyzed because 2 participants never initiated study drug.
Measure: Number (95% Confidence Interval); unit: Events per 100 patient-years
Arm/Group | Inosine | Placebo
Number analyzed (Participants) | 147 | 149
Events per 100 patient-years | 354.05 [330.18 to 379.64] | 327.73 [305.76 to 351.29]
Statistical Analysis 1: Comparison: Inosine vs Placebo; Test type: Other; p = 0.124, Poisson Regression; Rate Ratio = 1.080, 95% CI 2-sided [0.979 to 1.192]

3. Secondary Outcome: Percentage Developing Adverse Effects
Description: Safety of oral inosine titrated to elevate trough serum urate to 7.1 - 8.0 mg/dL will be evaluated by comparing active vs. placebo treatment with respect to the percentage of subjects experiencing individual types of AE, as classified by Medical Dictionary for Regulatory Activities (MedDRA) preferred term and system organ class.
Time Frame: two years
Population: Only 147 of 149 participants in the inosine group were analyzed because 2 participants never initiated study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Inosine | Placebo
Number analyzed (Participants) | 147 | 149
Participants | 129 | 137
Statistical Analysis 1: Comparison: Inosine vs Placebo; Test type: Other; p = 0.004, Poisson Regression; Rate Ratio = 1.154, 95% CI 2-sided [1.046 to 1.273]

4. Secondary Outcome: Percentage of Subjects Tolerant of the Treatment
Description: Tolerability of a treatment will be defined as a percentage of all subjects in a treatment group who are tolerant of the treatment at 12 weeks (short-term tolerability) and 24 months (long-term tolerability). A subject who is tolerant of treatment will be defined as one who remains on-study and on the assigned treatment without one or more dose reductions lasting more than 4 weeks cumulative due to AEs. A treatment will be declared tolerable if the percentage who are tolerant is significantly greater than 50% by one-tailed testing at p < 0.05.
Time Frame: three months; two years
Population: Only 147 of 149 participants in the inosine group were analyzed because 2 participants never initiated study drug.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Inosine | Placebo
Number analyzed (Participants) | 147 | 149
percentage of subjects
  12 weeks | 93.2 [87.7 to 96.3] | 98.7 [94.7 to 99.7]
  12 months | 76.1 [68.3 to 82.2] | 91.3 [85.4 to 94.8]
  24 months | 50.3 [39.2 to 60.5] | 70.8 [60.8 to 78.7]
Statistical Analysis 1: Comparison: Inosine vs Placebo; Test type: Other; p = 0.002, Log Rank

5. Secondary Outcome: Percentage of Participants Developing Disability Warranting Dopaminergic Therapy Over Time
Description: The percentage of participants with disability warranting the initiation of dopaminergic therapy in each treatment group at time from baseline visit (in 180 day increments).
Time Frame: two years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Inosine | Placebo
Number analyzed (Participants) | 149 | 149
percentage of participants
  0 Days | 0 [0 to 0] | 0 [0 to 0]
  180 Days | 30.81 [23.93 to 39.11] | 32.42 [25.53 to 40.61]
  360 Days | 59.01 [50.99 to 67.21] | 56.32 [48.50 to 64.44]
  540 Days | 72.21 [64.16 to 79.77] | 78.55 [71.12 to 85.16]
  720 Days | 84.57 [75.66 to 91.62] | 88.27 [81.29 to 93.54]
Statistical Analysis 1: Comparison: Inosine vs Placebo; Test type: Other; p = 0.497, Log Rank

6. Secondary Outcome: Clinical Efficacy: Rate of Change in Parkinson's Disease Questionnaire - 39 Item Version (PDQ-39) Scale
Description: Rate of change in Parkinson's Disease Questionnaire - 39 item version (PDQ-39) scale points (over the time between baseline visit and final visit on study drug) will be assessed for subjects in each treatment group. The PDQ-39 asks 39 questions organized over eight domains (scales): mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognition (4 items), communication (3 items), and bodily discomfort (3 items). Each item has five possible ordinal responses, from never to always, depending on frequency of the symptom over the preceding month. The eight scales' scores are generated by Likert's method of summated ratings and then transformed to a single figure that ranges from 0 to 100. Higher scores are associated with more symptoms.
Time Frame: two years
Measure: Mean (95% Confidence Interval); unit: score per year
Arm/Group | Inosine | Placebo
Number analyzed (Participants) | 149 | 149
score per year | 0.686 [0.094 to 1.278] | 0.756 [0.197 to 1.314]
Statistical Analysis 1: Comparison: Inosine vs Placebo; Test type: Other; p = 0.856, Mixed Models Analysis; Slope = -0.070, 95% CI 2-sided [-0.825 to 0.685], Standard Error of Mean 0.385

7. Secondary Outcome: Clinical Efficacy: Rate of Change in Quality of Life in Neurological Disorders (Neuro-QOL)
Description: Rate of change in Quality of Life in Neurological Disorders (Neuro-QOL) scale points (over the time between baseline visit and final visit on study drug) will be assessed for subjects in each treatment group. Neuro-QOL is a set of patient-reported outcome (PRO) measures that assess health-related quality of life (HRQoL) of people with neurological disorders. It comprises 17 domains of HRQL covering physical, psychological and social health. Domains tested include anxiety, cognitive function, communication, depression, emotional and behavioral dyscontrol, fatigue, lower extremity function- mobility, positive affect and well- being, stigma, upper extremity function- fine motor and ADL, sleep disturbance, satisfaction with social roles and activities, and ability to participate in social roles and activities. Higher raw scores are associated with more of the concept being measured. All scales range from 8 to 40 except for Positive Affect and Well-Being which ranges from 9 to 45.
Time Frame: two years
Measure: Mean (95% Confidence Interval); unit: score per year
Arm/Group | Inosine | Placebo
Number analyzed (Participants) | 149 | 149
score per year
  Anxiety | -0.397 [-0.757 to -0.037] | -0.473 [-0.818 to -0.129]
  Cognitive Function | 0.014 [-0.300 to 0.328] | -0.282 [-0.579 to 0.016]
  Communication | 0.055 [-0.106 to 0.215] | -0.201 [-0.353 to -0.049]
  Emotional and Behavioral Dyscontrol | -0.229 [-0.505 to 0.047] | -0.324 [-0.589 to -0.058]
  Fatigue | -0.049 [-0.482 to 0.383] | -0.040 [-0.455 to 0.375]
  Lower Extremity Function | -0.092 [-0.288 to 0.104] | -0.261 [-0.449 to -0.074]
  Positive Affect and Well-Being | -0.240 [-0.683 to 0.202] | 0.094 [-0.326 to 0.514]
  Stigma | -0.060 [-0.266 to 0.147] | 0.021 [-0.176 to 0.217]
  Upper Extremity Function | -0.026 [-0.243 to 0.191] | -0.238 [-0.446 to -0.030]
  Sleep Disturbance | 0.091 [-0.208 to 0.391] | 0.020 [-0.266 to 0.305]
  Satisfaction with Social Roles and Activities | -0.387 [-0.824 to 0.049] | -0.381 [-0.796 to 0.033]
  Participation in Social Roles and Activities | -0.382 [-0.883 to 0.118] | -0.130 [-0.611 to 0.352]
Statistical Analysis 1: Comparison: Inosine vs Placebo; Anxiety; Test type: Other; p = 0.736, Mixed Models Analysis; Slope = 0.076, 95% CI 2-sided [-0.368 to 0.521], Standard Error of Mean 0.226
Statistical Analysis 2: Comparison: Inosine vs Placebo; Cognitive Function; Test type: Other; p = 0.167, Mixed Models Analysis; Slope = 0.295, 95% CI 2-sided [-0.124 to 0.714], Standard Error of Mean 0.213
Statistical Analysis 3: Comparison: Inosine vs Placebo; Communication; Test type: Other; p = 0.022, Mixed Models Analysis; Slope = 0.256, 95% CI 2-sided [0.038 to 0.474], Standard Error of Mean 0.111
Statistical Analysis 4: Comparison: Inosine vs Placebo; Emotional and Behavioral Dyscontrol; Test type: Other; p = 0.584, Mixed Models Analysis; Slope = 0.095, 95% CI 2-sided [-0.245 to 0.435], Standard Error of Mean 0.173
Statistical Analysis 5: Comparison: Inosine vs Placebo; Fatigue; Test type: Other; p = 0.973, Mixed Models Analysis; Slope = -0.010, 95% CI 2-sided [-0.560 to 0.541], Standard Error of Mean 0.280
Statistical Analysis 6: Comparison: Inosine vs Placebo; Lower Extremity Function; Test type: Other; p = 0.214, Mixed Models Analysis; Slope = 0.169, 95% CI 2-sided [-0.098 to 0.437], Standard Error of Mean 0.136
Statistical Analysis 7: Comparison: Inosine vs Placebo; Positive Affect and Well-Being; Test type: Other; p = 0.271, Mixed Models Analysis; Slope = -0.334, 95% CI 2-sided [-0.931 to 0.262], Standard Error of Mean 0.304
Statistical Analysis 8: Comparison: Inosine vs Placebo; Stigma; Test type: Other; p = 0.566, Mixed Models Analysis; Slope = -0.080, 95% CI 2-sided [-0.355 to 0.194], Standard Error of Mean 0.140
Statistical Analysis 9: Comparison: Inosine vs Placebo; Upper Extremity Function; Test type: Other; p = 0.130, Mixed Models Analysis; Slope = 0.212, 95% CI 2-sided [-0.063 to 0.487], Standard Error of Mean 0.140
Statistical Analysis 10: Comparison: Inosine vs Placebo; Sleep Disturbance; Test type: Other; p = 0.723, Mixed Models Analysis; Slope = 0.072, 95% CI 2-sided [-0.325 to 0.468], Standard Error of Mean 0.202
Statistical Analysis 11: Comparison: Inosine vs Placebo; Satisfaction with Social Roles and Activities; Test type: Other; p = 0.984, Mixed Models Analysis; Slope = -0.006, 95% CI 2-sided [-0.592 to 0.579], Standard Error of Mean 0.298
Statistical Analysis 12: Comparison: Inosine vs Placebo; Participation in Social Roles and Activities; Test type: Other; p = 0.426, Mixed Models Analysis; Slope = -0.253, 95% CI 2-sided [-0.877 to 0.371], Standard Error of Mean 0.317

8. Secondary Outcome: Clinical Efficacy: Rate of Change in Quality of Life in Neurological Disorders (Neuro-QOL) Depression Module
Description: Rate of change in Quality of Life in Neurological Disorders (Neuro-QOL) depression module scale points (over the time between baseline visit and final visit on study drug) will be assessed for subjects in each treatment group. Neuro-QOL is a set of patient-reported outcome (PRO) measures that assess health-related quality of life (HRQoL) of people with neurological disorders. Higher raw scores are associated with more of the concept being measured. The depression module score ranges from 8 to 40.
Time Frame: two years
Measure: Mean (95% Confidence Interval); unit: score per year
Arm/Group | Inosine | Placebo
Number analyzed (Participants) | 149 | 149
score per year | -0.023 [-0.234 to 0.188] | 0.083 [-0.114 to 0.280]
Statistical Analysis 1: Comparison: Inosine vs Placebo; Test type: Other; p = 0.454, Mixed Models Analysis; Slope = -0.106, 95% CI 2-sided [-0.382 to 0.171], Standard Error of Mean 0.141

9. Secondary Outcome: Clinical Efficacy: Rate of Change in Schwab and England Scale
Description: Rate of change in percentage points on the Schwab and England scale for functional disability (over the time between baseline visit and final visit on study drug) will be assessed for subjects in each treatment group. The Schwab and England scale is a Site Investigator and subject assessment of the subject's level of independence. The subject will be scored on a percentage scale reflective of his/her ability to perform acts of daily living. Printed scores with associated descriptors range from 0% to 100% in increments of 5%, with higher percentages associated with more independence. A score of 0% implies "vegetative functions such as swallowing, bladder and bowel functions are not functioning; bedridden". A score of 100% implies "subject has full ability and is completely independent; essentially normal".
Time Frame: two years
Measure: Mean (95% Confidence Interval); unit: score per year
Arm/Group | Inosine | Placebo
Number analyzed (Participants) | 149 | 149
score per year | -0.833 [-1.536 to -0.131] | -0.880 [-1.555 to -0.206]
Statistical Analysis 1: Comparison: Inosine vs Placebo; Test type: Other; p = 0.910, Mixed Models Analysis; Slope = 0.047, 95% CI 2-sided [-0.764 to 0.858], Standard Error of Mean 0.413

10. Secondary Outcome: Clinical Efficacy: Rate of Change in Montreal Cognitive Assessment (MoCA)
Description: Rate of change in points on the Montreal Cognitive Assessment (MoCA) scale (for cognition; over the time between baseline visit and final visit on study drug) will be assessed for subjects in each treatment group. The MoCA assesses attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Points are awarded for the correct completion of MoCA tasks. Scores for each task are summed for a total score (range 0-30). Higher scores indicate greater cognitive capacity.
Time Frame: two years
Measure: Mean (95% Confidence Interval); unit: score per year
Arm/Group | Inosine | Placebo
Number analyzed (Participants) | 149 | 149
score per year | 0.186 [-0.012 to 0.384] | 0.226 [0.040 to 0.412]
Statistical Analysis 1: Comparison: Inosine vs Placebo; Test type: Other; p = 0.758, Mixed Models Analysis; Slope = -0.040, 95% CI 2-sided [-0.295 to 0.215], Standard Error of Mean 0.130

11. Secondary Outcome: Symptomatic Effects
Description: Symptomatic effects will be estimated by changes in motor and other features (e.g., as assessed by short-term change in Movement Disorders Society Unified PD Rating Scale [MDS-UPDRS] I-III total score) during the first 3 months of wash-in at the start of period 1 and during the 3-month wash-out of period 2. The MDS-UPDRS includes ratings of non-motor experiences of daily living, motor experiences of daily living, and a motor examination. The MDS-UPDRS is assessed on a 5-point Likert scale ranging from 0 to 4 where higher scores imply worse features. Parts I-III contain 59 total questions (13 in Part I, 13 in Part II, and 33 in Part III). Total scores are calculated as simple sums of component items with mean imputation by Part if no more than 1, 2, or 7 items are missing for Parts I through III, respectively. Total scores may range from 0 to 236, with 0 meaning no symptoms and 236 meaning worse symptoms.
Time Frame: three months (after both initiation and discontinuation of study drug)
Measure: Mean (95% Confidence Interval); unit: score per period
Arm/Group | Inosine | Placebo
Number analyzed (Participants) | 149 | 149
score per period
  Period 1: BL to V03 | -1.509 [-2.656 to -0.362] | -1.301 [-2.433 to -0.169]
  Period 2: V10 to SV | -2.729 [-7.746 to 2.289] | -0.328 [-4.762 to 4.105]
Statistical Analysis 1: Comparison: Inosine vs Placebo; BL to V01; Test type: Other; p = 0.796, Mixed Models Analysis; Slope = -0.208, 95% CI 2-sided [-1.783 to 1.367], Standard Error of Mean 0.803
Statistical Analysis 2: Comparison: Inosine vs Placebo; V10 to SV; Test type: Other; p = 0.486, Mixed Models Analysis; Slope = -2.400, 95% CI 2-sided [-9.156 to 4.355], Standard Error of Mean 3.443

ADVERSE EVENTS:
Time Frame: 27 months
Description: Only 147 of 149 participants in the inosine group were analyzed because 2 participants never initiated study drug.
Arm/Group | Inosine | Placebo
All-Cause Mortality (participants affected / at risk) | 1/147 | 0/149
Serious Adverse Events (participants affected / at risk) | 16/147 | 21/149
Other Adverse Events (participants affected / at risk) | 125/147 | 135/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inosine (N=147) | Placebo (N=149)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2)
Death (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Extradural abscess (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (3)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 6 (6) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Testicular mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 2 (2)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inosine (N=147) | Placebo (N=149)
Constipation (Gastrointestinal disorders) | 7 (7) | 16 (16)
Diarrhoea (Gastrointestinal disorders) | 9 (11) | 9 (12)
Nausea (Gastrointestinal disorders) | 22 (25) | 20 (31)
Fatigue (General disorders) | 8 (9) | 11 (11)
Nasopharyngitis (Infections and infestations) | 12 (14) | 10 (13)
Sinusitis (Infections and infestations) | 10 (11) | 7 (9)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 13 (16)
Urinary tract infection (Infections and infestations) | 17 (24) | 10 (16)
Blood creatinine increased (Investigations) | 13 (13) | 3 (3)
Crystal urine present (Investigations) | 8 (9) | 7 (9)
Mean cell volume increased (Investigations) | 12 (13) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 13 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (19) | 10 (12)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 (10) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9) | 21 (25)
Dizziness (Nervous system disorders) | 14 (16) | 16 (22)
Headache (Nervous system disorders) | 8 (9) | 14 (16)
Somnolence (Nervous system disorders) | 4 (4) | 8 (9)
Insomnia (Psychiatric disorders) | 9 (9) | 6 (6)
Haematuria (Renal and urinary disorders) | 13 (13) | 12 (12)
Nephrolithiasis (Renal and urinary disorders) | 12 (12) | 4 (4)
Proteinuria (Renal and urinary disorders) | 9 (9) | 12 (14)

LIMITATIONS AND CAVEATS:
A prespecified interim analysis determined futility for demonstrating the hypothesized inosine effect of a slower rate of change in the primary outcome and prompted early completion of the trial after an average study drug exposure of 17 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT02642393/SAP_000.pdf
  • Study Protocol (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT02642393/Prot_001.pdf